CLINICAL TRIAL: NCT03764423
Title: Health Effects of Salmon Fishmeal in Humans With Impaired Glucose Tolerance
Brief Title: Health Effects of Salmon Fishmeal in Humans
Acronym: FishMeal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Kirsten Holven, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 901420
Record Dates: First submitted 2018-06-29; First posted 2018-12-05 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Fish Proteins; microcrystalline cellulose; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salmon fishmeal (Experimental): 7,5 g fishmeal and 7,5 g microcrytalline cellulose per day in capsules by mounth for 8 weeks
  Interventions: Dietary Supplement: Salmon fishmeal
- Microcrystalline cellulose (Placebo Comparator): 7,5 g microcrystalline cellulose per day in capsules by mounth for 8 weeks
  Interventions: Dietary Supplement: Microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Salmon fishmeal — Salmon fishmeal with high protein content
  Other Names: Fish protein
  Arms: Salmon fishmeal
Dietary Supplement: Microcrystalline cellulose — Microcrystalline cellulose contain no energy and is less fermented in the gut than other dietary fibers.
  Other Names: Cellulose
  Arms: Microcrystalline cellulose

SUMMARY:
Diabetes contributes significantly to the burden of disease in Norway and cardiovascular disease is the main cause of mortality.

Both lean and fatty fish are shown to have beneficial health effects. In addition to omega-3 fatty acids, fish contain potential health-promoting components such as taurine, vitamin D, vitamin B12, iodine, selenium and more unspecified components such as bioactive peptides. With the expected growth in the aquaculture sector, more protein-rich by-products will become available.

The overall aim of this project is to investigate the health beneficial effects of fish protein in the form of salmon fishmeal in a human intervention study with regard to metabolic risk markers.

We will include subjects with impaired glucose tolerance to a randomized controlled parallel study. The subjects will receive capsules with fishmeal or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose ≥ 5.6 mmol/l or
* Plasma glucose ≥ 6.5 mmol/l 2h after an OGTT or
* HbA1c ≥ 5.8 %

Exclusion criteria:

* Diabetes (defined as p-glucose ≥ 7.0 mmol/l p-glucose ≥11,1 mmol/l 2h after OGTT or HbA1c ≥ 6.5 %)
* High fish intake (> 450 gram/week) or fish allergy
* Age-related elevated blood pressure (≥ 70 år: ≥ 180/110 mmHg, > 40-70: ≥ 170/100 mmHg and ≤ 40 år: ≥ 160/100 mmHg)
* Use of prescription medicines related to diabetes, inflammation, systemic use of corticosteroids.
* Non-stable use of lipid lowering drugs, thyroxine, blood pressure lowering drugs, drugs affecting appetite, dietary supplements (including n-3)
* High intake of protein supplements powder
* Pregnancy
* Planning pregnancy or changes in body weight

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
2 hour postprandial blood glucose concentration | Change in 2 hour blood glucose concentration from baseline and after 8 weeks between groups
  Glucose concentration measured before and after a standard glucose tolerance test at baseline and after 8 weeks
Fasting blood glucose concentration | Change in blood glucose concentration from baseline and after 8 weeks between groups
  Measured at baseline and after 8 weeks.

SECONDARY OUTCOMES:
Blood concentration of insulin | Changes in blood insulin concentration from baseline and after 8 weeks between groups
  Blood concentration measured fasting and 2 hours after an oral glucose tolerance test
HOMA-IR | Changes in HOMAR-IR from baseline and after 8 weeks between groups
  Blood concentration of insulin x blood concentration of glucose will be used to calculate HOMAR-IR fasting and 2 hours after an oral glucose tolerance test
Blood concentration of HbA1c | Changes in blood HbA1c concentration from baseline and after 8 weeks between groups
  Blood concentration measured fasting
Blood concentration of incretins (i.e. GLP-1) | Changes in blood glucose concentration of increstins from baseline and after 8 weeks between groups
  Blood concentration of incretins measured fasting and 2 hours after oral glucose tolerance test

OTHER OUTCOMES:
Markers related to lipid metabolism | Changes in blood concentrations of markers related to lipid metabolism from baseline and after 8 weeks intervensjon
  Blood concentrations of i.e. triglycerides, total-, LDL- and HDL- cholesterol, free fatty acids and lipoprotein subclasses (lipidomics)
Markers related to low grade inflammation, including changes in genes expression level in peripheral blood mononuclear cell (PBMCs) in circulation | Changes in blood concentrations of markers related to inflammation from baseline and after 8 weeks between groups
  Blood concentrations of i.e. CRP, IL-6
Markers related to appetite | Changes in blood concentrations of markers related to appetite from baseline and after 8 weeks between groups
  Blood concentrations of gut hormones, i.e. PYY, amylin, leptin
Changes in PBMC wholegenome transcriptome and untargeted metabolomics | Changes in blood concentration of PBMC wholegenome transcriptome and untargeted metabolomics from baseline and after 8 weeks whithin and between groups
  Blood or urine transcriptome and metabolomics
Changes in markers related to gut microbiota | Changes in markers related to gut microbiota between groups from baseline and after 8 weeks intervensjon
  Faecal short-chain fatty acids, bacteria type and diversity
Changes in blood concentration of micronutrients related to fishintake | Changes in blood concentrations of micronutrients related to fishintake between groups from baseline and after 8 weeks intervensjon
  Blood concentrations of i.e. vitamin D, Zn, Se and iodine
Changes in blood concentration of amino acids | Changes in blood concentrations of amino acids between groups postprandially, and between baseline and 8 weeks of intervention
  Blood concentrations of different aminoacids such as i.e valine, isoleucine, leucine
Body weight | Change between groups from baseline and after 8 weeks intervensjon will be calculated
  Bodyweight (kg) will be used to calculate i.e BMI (kg/m2)
Height | Change between groups from baseline and after 8 weeks intervensjon will be calculated
  Height (m) will be used to calculate i.e. BMI (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Holven, Professor, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Post Box 1046, Blindern, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hustad KS, Ottestad I, Olsen T, Saether T, Ulven SM, Holven KB. Salmon fish protein supplement increases serum vitamin B12 and selenium concentrations: secondary analysis of a randomised controlled trial. Eur J Nutr. 2022 Sep;61(6):3085-3093. doi: 10.1007/s00394-022-02857-4. Epub 2022 Apr 1. PMID 35362766